CLINICAL TRIAL: NCT06474078
Title: An Open-Label Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of Tofacitinib in Patients With Stevens-Johnson Syndrome (SJS) and Toxic Epidermal Necrolysis (TEN)
Brief Title: Study To Evaluate The Efficacy Of Tofacitinib In Patients With SJS/TEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun Bing Chen, Principal Investigator, Clinical Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202102411A3
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolysis
Keywords: JAK/STAT Pathway; Stevens-Johnson Syndrome; Toxic Epidermal Necrolysis; JAK1/3 inhibitor; Tofacitinib
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofacitinib treatment (Experimental): 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do serum granulysin concentration and peripheral blood mononuclear spherical granulysin expression analysis
  4. Tofacitinib administration: The experimental group received tofacitinib 5mg-10mg, twice daily, for the first week; and maintained tofacitinib 5mg-10mg, daily, for the second week.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Dosage/Frequency: 5mg - 10mg, oral, twice daily
  Other Names: XELJANZ

SUMMARY:
The goal of this study is to evaluate the effect of tofacitinib in patients with Stevens-Johnson Syndrome (SJS) and Toxic Epidermal Necrolysis (TEN). The primary outcome of the study is the time to complete re-epithelialization. The secondary outcomes are to determine mortality, length of hospitalization, adverse events, the time to beginning of epithelization, the time to halting of progression of SJS/TEN, ocular complications, and infections.

DETAILED DESCRIPTION:
Stevens-Johnson syndrome (SJS) and toxic epidermal necrolysis (TEN) belong to life-threatening severe cutaneous adverse drug reactions. SJS/TEN is classified by the extent of the detachment over the total body-surface area: SJS (<10%), SJS-TEN overlap (10%-30%), and TEN (>30%). TEN has the highest mortality (30-35%); SJS and transitional forms correspond to the same syndrome, but with less extensive skin detachment and a lower mortality (5-15%). Currently, there is still no conclusive effective immunomodulator treatment for SJS/TEN. And, there is still a clinical unmet need for the treatment of SJS/TEN.

According to our past research reports, interleukin-15 (IL-15) plays an important role in SJS/TEN, which is related to disease severity and mortality. Janus kinase (JAK) inhibitors can inhibit the downstream JAK to inhibit the production and transmission of inflammatory cytokines, as a treatment for severe skin drug hypersensitivity reactions. Tofacitinib, a JAK1/3 inhibitor, is an intervention known to effectively treat several inflammatory diseases including rheumatoid arthritis, psoriatic arthritis, and ulcerative colitis. Notably, a recent study identified a potential therapeutic target with JAK-STAT pathway in a patient with recalcitrant and refractory drug rash with eosinophilia and systemic symptoms (DRESS). Based the current evidence, a targeting therapy to IL-15 by tofacitinib treatment are suggesting likely to be effective in treating SJS/TEN.

This is an "open label" study, all patients enrolled in the study will receive the active medication; meaning that there will not be a placebo or control group. The aims of this project are (1) to investigate the effect of tofacitinib treatment for SJS/TEN patients, including healing time, mortality rate, adverse events, beginning of re-epithelialization time, internal organ recovery time, and ocular complications, and (2) to investigate the molecular mechanism of SJS/TEN after tofacitinib treatment through collection of timed samples to include DNA, RNA, PBMCs, blister cells and supernatant and skin tissue.

The primary outcome of the study is the time to complete re-epithelialization as defined by complete absence of erosion on the skin. The secondary outcomes are to determine the time to beginning of epithelization (defined as the time to start re-epithelialization of the erosions on the skin and mucosa), the time to halting of progression of SJS/TEN (considered significant progression if there are any new blistering lesions or any new detached or detachable skin), mortality, length of hospitalization, ocular complications, infections, and adverse events. The investigators also determine the molecular and cellular mechanisms of SJS/TEN through collection of timed samples to include DNA, RNA, PBMCs, blister cells and supernatant and skin tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign inform consent form
2. Subject has been diagnosed with Stevens-Johnson syndrome or toxic epidermal necrolysis by at least two dermatologists.
3. Male or female aged over 20 years old and under 90 years old.

Exclusion Criteria:

1. Subject or legally authorized representative is not willing to provide informed consent.
2. Women who are pregnant or breastfeeding
3. Subject has an active, untreated, or serious infectious disease that is ineffective in treatment, such as sepsis.
4. Subject suffers from severe life-threatening cardiac arrhythmia, such as ventricular tachycardia, have had myocardial infarction (myocardial infarction), severe hypertension that has not responded to treatment within the past week, or other cardiologist diagnosed severe cardiovascular disease
5. Subject has active viral hepatitis
6. Subject has active tuberculosis
7. Subject received live vaccination during the illness

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Bing Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SCAR patients were enrolled in the clinical trial from 2022/08/01 to 2025/04/15 at Chang Gung Memorial Hospital in Taiwan.
Pre-assignment Details: SJS/TEN (n=20)
Groups:
- Tofacitinib Treatment: 1. Meet the conditions of inclusion and exclusion, seek the consent of the patient
  2. Fill out the case report form
  3. Blood test and physiological assessment, and do serum granulysin concentration and peripheral blood mononuclear spherical granulysin expression analysis
  4. Tofacitinib administration: The experimental group received tofacitinib 5mg-10mg, twice daily, for the first week; and maintained tofacitinib 5mg-10mg, daily, for the second week.
  Tofacitinib: Dosage/Frequency: 5mg - 10mg, oral, twice daily
Period: Overall Study
Arm/Group | Tofacitinib Treatment
Started | 20 (SJS/TEN (n=20))
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We totally recruited 20 SJS/TEN participants to analyze.
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 20
Blister/erosion [Count of Participants; unit: Participants] | 14
Fever, >38℃ [Count of Participants; unit: Participants] | 11
Atypical target lesion [Count of Participants; unit: Participants] | 11
GPT, > 82 U/L [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Skin Healing Time, Day, Medium [Full Range]
Description: Healing was defined as complete re-epithelialization (i.e., the complete absence of erosions). We recorded the time taken by the skin to heal.
Time Frame: days
Population: We determined if the enrolled participants had SJS/TEN using the criteria and histopathological examinations.
Measure: Median (Full Range); unit: days
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 20
days | 10.0 [6 to 15]

2. Primary Outcome: Complete Skin Healing Time, Day, Mean [Full Range]
Description: as for outcome 1
Time Frame: days
Population: We determined if the enrolled participants had SJS/TEN using the criteria and histopathological examinations.
Measure: Mean (Full Range); unit: days
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 20
days | 10.1 [6 to 15]

3. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization and Duration of hospitalization days
Time Frame: Duration of hospital stay up to 3 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Tofacitinib Treatment: Duration of hospital stay after tofacitinib treatment.
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 20
days | 22.4 (15.6)

4. Secondary Outcome: Mortality
Description: Number of participants with mortality at 30 days, 3 months and 1 year. Mortality monitoring is considered for the underlying SJS/TEN disease.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Treatment: Observed mortality=0 %
Arm/Group | Tofacitinib Treatment
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were assessed three weeks to three months. Moreover, all-cause mortality was assessed up to 1 year.
Description: AEs surveillance began at the initiation of tofacitinib and continued through three weeks after the final dose, serving as the predefined safety endpoint.
  The duration of clinical and laboratory monitoring as well as AEs evaluation ranged from 1 to 3 months.
  AEs monitoring pertains to post-tofacitinib treatment.
  Serious and other (not including serious) adverse events were assessed three weeks to three months.
  Moreover, all-cause mortality was assessed up to 1 year.
Arm/Group | Tofacitinib Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Treatment (N=20)
Abnormal liver function (Hepatobiliary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT06474078/Prot_SAP_000.pdf